CLINICAL TRIAL: NCT02230254
Title: PE PREMIER China: A Prospective, Multicenter Trial to Assess the Promus PREMIER Everolimus-Eluting Platinum Chromium Coronary Stent System for the Treatment of Atherosclerotic Lesion(s)
Brief Title: PE PREMIER CHINA CLINICAL TRIAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2323
Record Dates: First submitted 2014-08-20; First posted 2014-09-03 (Estimated); Results first posted 2022-05-12 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-02

CONDITIONS: Atherosclerosis
Keywords: Coronary Artery Disease
MeSH Terms: conditions — Atherosclerosis; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PROMUS POREMIER stent (Experimental): Single-arm treatment group receiving interventional PROMUS PRIMIER study stent
  Interventions: Device: Percutaneous coronary intervention PROMUS PREMIER

INTERVENTIONS:
Device: Percutaneous coronary intervention PROMUS PREMIER — PROMUS PREMIER

SUMMARY:
PE PREMIER China: A Prospective, Multicenter Trial to Assess the Promus PREMIERTM Everolimus-Eluting Platinum Chromium Coronary Stent System for the Treatment of Atherosclerotic Lesion(s)

DETAILED DESCRIPTION:
To evaluate clinical and peri-procedural angiographic outcomes for the Promus PREMIERTM Everolimus-Eluting Platinum Chromium Coronary Stent System in the treatment of subjects with atherosclerotic lesion(s) ≤34 mm in length (by visual estimate) in native coronary arteries ≥2.25 mm to ≤4.0 mm in diameter (by visual estimate)

ELIGIBILITY:
Inclusion Criteria:

* Clinical Inclusion (CI) Criteria

CI1. Subject must be at least 18 -75 years of age

CI2. Subject (or legal guardian) understands the trial requirements and the treatment procedures and provides written informed consent before any trial-specific tests or procedures are performed

CI3. Subject is eligible for percutaneous coronary intervention (PCI)

CI4. Subject has symptomatic coronary artery disease with objective evidence of ischemia or silent ischemia

CI5. Subject is an acceptable candidate for coronary artery bypass grafting (CABG)

CI6. Subject is willing to comply with all protocol-required follow-up evaluation

CI7. Subject has a left ventricular ejection fraction (LVEF) >30% as measured within 60 days prior to enrollment

* Angiographic Inclusion (AI) Criteria (visual estimate)

AI1. Target lesion(s) must be located in a native coronary artery with a visually estimated reference vessel diameter (RVD) ≥2.25 mm and ≤4.0 mm

AI2. Target lesion(s) length must be ≤34 mm ( Target lesion(s) length must be ≤28 mm for reference vessel diameter (RVD) = 2.25 mm Target lesion(s)) (by visual estimate)

AI3. Target lesion(s) must have visually estimated stenosis ≥50% and <100% with thrombolysis in Myocardial Infarction (TIMI) flow >1 and one of the following (stenosis ≥70%, abnormal fractional flow reserve (FFR), abnormal stress test or imaging stress test, or elevated biomarkers) prior to procedure

AI4. Coronary anatomy is likely to allow delivery of a study device to the target lesions(s)

AI5. The first lesion treated must be successfully pre-dilated/pretreated Note: Successful pre-dilatation/pretreatment refers to dilatation with a balloon catheter of appropriate length and diameter, or pretreatment with/or rotational coronary atherectomy, or cutting/scoring balloon with no greater than 50% residual stenosis and no dissection greater than National Heart, Lung, Blood Institute (NHLBI) type C.

Exclusion Criteria:

* Clinical Exclusion (CE) Criteria

CE1. Subject has clinical symptoms and/or electrocardiogram (ECG) changes consistent with Acute MI (include STEMI and Non- STEMI ) within 1 week

CE2. Subject has cardiogenic shock, hemodynamic instability requiring inotropic or mechanical circulatory support, intractable ventricular arrhythmias, or ongoing intractable angina

CE3. Subject has received an organ transplant or is on a waiting list for an organ transplant

CE4. Subject is receiving or scheduled to receive chemotherapy within 30 days before or after the index procedure

CE5. Planned PCI (including staged procedures) or CABG after the index procedure

CE6. Subject previously treated at any time with intravascular brachytherapy

CE7. Subject has a known allergy to contrast (that cannot be adequately pre-medicated) and/or the trial stent system or protocol-required concomitant medications (e.g., platinum, platinum-chromium alloy, stainless steel, everolimus or structurally related compounds, polymer or individual components, Clopidogrel , or aspirin)

CE8. Subject has one of the following (as assessed prior to the index procedure):

* Other serious medical illness (e.g., cancer, congestive heart failure) with estimated life expectancy of less than 12 months
* Current problems with substance abuse (e.g., alcohol, cocaine, heroin, etc.)
* Planned procedure that may cause non-compliance with the protocol or confound data interpretation

CE9. Subject is receiving chronic (≥72 hours) anticoagulation therapy (i.e., heparin, coumadin) for indications other than acute coronary syndrome

CE10. Subject with out of range complete blood count (CBC) values that are determined by the study physician to be clinically significant.

CE11. Subject has documented or suspected liver disease, including laboratory evidence of hepatitis

CE12. Subject is on dialysis or has baseline serum creatinine level >2.0 mg/dL (177µmol/L)

CE13. Subject has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions

CE14. Subject has had a history of cerebrovascular accident (CVA) or transient ischemic attack (TIA) within the past 6 months

CE15. Subject has an active peptic ulcer or active gastrointestinal (GI) bleeding

CE16. Subject has signs or symptoms of active heart failure (i.e., NYHA class IV) at the time of the index procedure

CE17. Subject is participating in another investigational drug or device clinical trial that has not reached its primary endpoint

CE18. Subject intends to participate in another investigational drug or device clinical trial within 12 months after the index procedure

CE19. Subject with known intention to procreate within 12 months after the index procedure (women of child-bearing potential who are sexually active must agree to use a reliable method of contraception from the time of screening through 12 months after the index procedure)

CE20. Subject is a woman who is pregnant or nursing (a pregnancy test must be performed within 7 days prior to the index procedure in women of child-bearing potential)

CE21.Target vessel has been treated with any type of PCI (e.g., balloon angioplasty, stent, cutting balloon, atherectomy) within 12 months prior to the index procedure

* Angiographic Exclusion (AE) Criteria (visual estimate)

AE1. Planned treatment of more than 3 lesions.

AE2. Planned treatment of lesions in more than 2 major epicardial vessels

AE3. Planned treatment of a single lesion with more than 1 stent

AE4. Subject has 2 target lesions in the same vessel that are separated by less than 20 mm (by visual estimate)

AE5. Target lesion(s) is located in the left main

AE6. Target lesion(s) is located within 3 mm of the origin of the left anterior descending (LAD) coronary artery or left circumflex (LCx) coronary artery by visual estimate.

AE7. Target lesion(s) is located within a saphenous vein graft or an arterial graft

AE8. Target lesion(s) will be accessed via a saphenous vein graft or arterial graft

AE9. Target lesion(s) with a TIMI flow 0 (total occlusion) or TIMI flow 1 prior to guide wire crossing

AE10. Target lesion(s) treated during the index procedure that involves a complex bifurcation (e.g., bifurcation lesion requiring treatment with more than 1 stent)

AE11. Target lesion(s) is restenotic from a previous stent implantation or study stent would overlap with a previous stent

AE12. Subject has unprotected left main coronary artery disease (>50% diameter stenosis)

AE13. Subject has been treated with any type of PCI (i.e., balloon angioplasty, stent, cutting balloon atherectomy) within 24 hours prior to the index procedure

AE14. Thrombus, or possible thrombus, present in the target vessel (by visual estimate)

AE15. Excessive tortuosity proximal to or within the lesion

AE16. Excessive angulation proximal to or within the lesion

AE17. Target lesion and/or the target vessel proximal to the target lesion is moderately to severely calcified by visual estimate

AE18. Involves a side branch ≥2.0 mm in diameter by visual estimate or a side branch <2.0 mm in diameter by visual estimate which requires treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2014-04-09 (Actual); Primary Completion 2014-06-22 (Actual); Study Completion 2015-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jian'an Wang, Doctor, Principal Investigator — 2nd affiliated hospital of Zhejiang University College of Medicine

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total Started: 101
Period: Overall Study
Arm/Group | PROMUS POREMIER Stent
Started | 101
Completed | 98
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | PROMUS POREMIER Stent
Number analyzed (Participants) | 101
Age, Continuous [Mean (Standard Deviation); unit: Year] | 61.47 (9.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 77

OUTCOME MEASURES:

1. Primary Outcome: Technical Success Rate
Description: Technical success rate, defined as successful delivery and deployment of the study stent to the target lesion, without balloon rupture or stent embolization, and post-procedure diameter stenosis of <30% assessed in 2 near-orthogonal projections with TIMI 3 flow in the target lesion, as visually assessed by the physician
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS POREMIER Stent
Number analyzed (Participants) | 101
percentage of participants | 99.1

2. Secondary Outcome: Target Lesion Revascularization (TLR) Rate
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day, at 30 days, 6months and 12months
Reporting Status: Not Posted

3. Secondary Outcome: Target Lesion Failure (TLF) Rate
Time Frame: as for outcome 2
Reporting Status: Not Posted

4. Secondary Outcome: Target Vessel Revascularization (TVR) Rate
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day, at 30 days, 6month and 12months
Reporting Status: Not Posted

5. Secondary Outcome: Target Vessel Failure (TVF) Rate
Time Frame: as for outcome 2
Reporting Status: Not Posted

6. Secondary Outcome: Myocardial Infarction (MI, Q-wave and Non-Q-wave) Rate
Time Frame: as for outcome 2
Reporting Status: Not Posted

7. Secondary Outcome: Cardiac Death Rate
Time Frame: as for outcome 2
Reporting Status: Not Posted

8. Secondary Outcome: Non-cardiac Death Rate
Time Frame: as for outcome 2
Reporting Status: Not Posted

9. Secondary Outcome: All Death Rate
Time Frame: as for outcome 2
Reporting Status: Not Posted

10. Secondary Outcome: Cardiac Death or MI Rate
Time Frame: as for outcome 2
Reporting Status: Not Posted

11. Secondary Outcome: All Death or MI Rate
Time Frame: as for outcome 2
Reporting Status: Not Posted

12. Secondary Outcome: All Death/MI/TVR Rate
Time Frame: as for outcome 2
Reporting Status: Not Posted

13. Secondary Outcome: Stent Thrombosis Rate (by Academic Research Consortium [ARC] Definitions)
Time Frame: as for outcome 2
Reporting Status: Not Posted

14. Secondary Outcome: Clinical Procedural Success Rate
Time Frame: as for outcome 2
Reporting Status: Not Posted

15. Secondary Outcome: In-stent and In-segment Percent Diameter Stenosis (%DS)
Time Frame: as for outcome 2
Reporting Status: Not Posted

16. Secondary Outcome: In-stent and In-segment Minimum Lumen Diameter (MLD)
Time Frame: as for outcome 2
Reporting Status: Not Posted

17. Secondary Outcome: Acute Gain
Description: as measured by angiographic core lab, change from baseline for target lesions
Time Frame: as for outcome 2
Reporting Status: Not Posted

18. Secondary Outcome: Longitudinal Stent Deformation (LSD) Rate
Time Frame: as for outcome 2
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | PROMUS POREMIER Stent
All-Cause Mortality (participants affected / at risk) | 0/101
Serious Adverse Events (participants affected / at risk) | 8/101
Other Adverse Events (participants affected / at risk) | 13/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PROMUS POREMIER Stent (N=101)
Angina pectoris (Cardiac disorders) | 3 (4)
Angina unstable (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PROMUS POREMIER Stent (N=101)
Angina pectoris (Cardiac disorders) | 9 (9)
Angina unstable (Cardiac disorders) | 1 (1)
Coronary artery dissection (Cardiac disorders) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes